CLINICAL TRIAL: NCT01129128
Title: 3-arm Randomized Controlled Trial Assessing the in Vivo Effect of an Echinacea Purpurea on Immune Markers in Adults
Brief Title: Three Arm Trial of Immune Effects of Echinacea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, James Taylor, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 10A1276
Record Dates: First submitted 2010-05-14; First posted 2010-05-24 (Estimated); Results first posted 2012-06-05 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Upper Respiratory Tract Infections
Keywords: Echinacea; immune modulation; prevention
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Echinacea preparation 1 (Active Comparator): Commercially available Echinacea purpurea product
  Interventions: Biological: Echinacea purpurea product
- Echinacea preparation 2 (Active Comparator): Commercially available Echinacea purpurea product
  Interventions: Biological: Echinacea purpurea product
- Placebo (Placebo Comparator): Inert liquid that is similar in appearance and taste to the active Echinacea products
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Echinacea purpurea product — 5 ml by mouth 3 times per day for 10 days
  Arms: Echinacea preparation 1
Biological: Echinacea purpurea product — 1 ml by mouth 3 times per day for 10 days
  Arms: Echinacea preparation 2
Biological: Placebo — either 5 ml or 1 ml by mouth three times per day for 10 days
  Arms: Placebo

SUMMARY:
The goal of this study is to determine if either of two, commercially available, Echinacea purpurea products stimulate the immune system. For the study, 60 healthy adults will be randomized to receive one of the two Echinacea purpurea products or placebo for 10 days. Blood will be drawn to assess immune markers just before beginning the study medication, during the 10 day course of medication and after completing the course of medication. It is postulated that adults receiving either of the Echinacea products will have evidence of immune stimulation and those receiving placebo will not.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult (based on a screening health questionnaire)
* Speaks and reads English.
* If female of child-bearing potential, willing to use contraception to prevent pregnancy during the study.
* No use of any medication (other than multivitamins, essential fatty acids, oral contraceptives and probiotics) for 2 weeks prior to first dose of study.
* Willing to abstain from ingesting edible mushrooms for 2 weeks prior and throughout study.
* Willing to eat less than 2 garlic cloves per day for 2 weeks prior and during the study period

Exclusion Criteria:

* Pregnancy or currently breastfeeding.
* History of autoimmune disease or immune disorders.
* History of asthma.
* History of allergic rhinitis.
* History of physician diagnosed eczema, psoriasis or other skin condition that could mask an Echinacea-induced rash.
* Known allergic reaction to Echinacea or related species, specifically ragweed (Ambrosia), chamomile (Matricaria), goldenrod (Solidago), and sunflower (Helianthus).
* Known allergic reaction to xylitol sweetener, glycerine, citric acid, or citrus fruits

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Taylor, MD, Principal Investigator — University of Washington
Locations (1):
- Bastyr University, Kenmore, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adult volunteers enrolled from May 2010 through March 2011
Groups:
- Commercially Available Echinacea Product #1 (5 ml/Dose): Echinacea purpurea product; 5 ml dose administered three times daily for 10 days
- Commercially Available Echinacea Product #2 (1 ml/Dose): Echinacea purpurea product; 1 ml dose administered three times daily for 10 days
Period: Overall Study
Arm/Group | Commercially Available Echinacea Product #1 (5 ml/Dose) | Commercially Available Echinacea Product #2 (1 ml/Dose) | Placebo
Started | 22 | 22 | 23
Completed | 19 | 18 | 19
Not Completed | 3 | 4 | 4
Not completed — Lost to Follow-up | 2 | 2 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 3
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Commercially Available Echinacea Product #1 (5 ml/Dose) | Commercially Available Echinacea Product #2 (1 ml/Dose) | Placebo | Total
Number analyzed (Participants) | 22 | 22 | 23 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 23 | 67
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34.1 (10.6) | 35.1 (13.5) | 28.2 (8.0) | 32.4 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 17 | 47
  Male | 6 | 8 | 6 | 20
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 23 | 67

OUTCOME MEASURES:

1. Primary Outcome: Peak Level of TNF Alpha
Description: Highest level of TNF alpha while taking study medication
Time Frame: 1-10 days after starting study medication
Population: Data analyzed on any participant who TNF alpha level was obtained on 1 or more days while on study medication.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Commercially Available Echinacea Product #1 (5 ml/Dose) | Commercially Available Echinacea Product #2 (1 ml/Dose) | Placebo
Number analyzed (Participants) | 22 | 22 | 22
pg/ml | 436 (510) | 1467 (2330) | 721 (1272)
Statistical Analysis 1: Comparison: Commercially Available Echinacea Product #1 (5 ml/Dose) vs Placebo; comparison of peak level of TNF alpha after controlling for baseline level. Based on data from 20 participants in a group, there was a power of 0.9 to detect a difference of 1000 pg/ml with a standard deviation of 700 pg/ml; Test type: Superiority or Other; p = 0.87, Regression, Linear; controlled for baseline levels and performed log transformation of TNF alpha levels to account for skewed distribution of values; Mean Difference (Final Values) = -173
Statistical Analysis 2: Comparison: Commercially Available Echinacea Product #2 (1 ml/Dose) vs Placebo; comparison of peak level of TNF alpha after controlling for baseline level. Based on data from 20 participants in a group, there was a power of .9 to detect a difference of 1000 pg/ml with a standard deviation of 700 pg/ml; Test type: Superiority or Other; p = 0.82, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 705

2. Secondary Outcome: Peak Level IL-6
Description: Highest level of IL-6 while taking study medication
Time Frame: 1-10 days after starting study medication
Population: Data analyzed on any participant who IL-6 level was obtained on 1 or more days while on study medication.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Commercially Available Echinacea Product #1 (5 ml/Dose) | Commercially Available Echinacea Product #2 (1 ml/Dose) | Placebo
Number analyzed (Participants) | 22 | 22 | 22
pg/ml | 16296 (37448) | 44901 (79868) | 28526 (61921)
Statistical Analysis 1: Comparison: Commercially Available Echinacea Product #1 (5 ml/Dose) vs Placebo; Test type: Superiority or Other; p = 0.82, Regression, Linear; controlled for baseline levels and performed log transformation of IL-6 levels to account for skewed distribution of values; Mean Difference (Final Values) = -15793
Statistical Analysis 2: Comparison: Commercially Available Echinacea Product #2 (1 ml/Dose) vs Placebo; Test type: Superiority or Other; p = 0.68, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 23472

3. Secondary Outcome: Peak Level Interferon Gamma
Description: Highest level of Interferon gamma while taking study medication
Time Frame: 1-10 days after starting study medication
Population: Data analyzed on any participant who Interferon gamma level was obtained on 1 or more days while on study medication.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Commercially Available Echinacea Product #1 (5 ml/Dose) | Commercially Available Echinacea Product #2 (1 ml/Dose) | Placebo
Number analyzed (Participants) | 22 | 22 | 22
pg/ml | 74 (122) | 146 (321) | 121 (292)
Statistical Analysis 1: Comparison: Commercially Available Echinacea Product #1 (5 ml/Dose) vs Placebo; Test type: Superiority or Other; p = 0.90, Regression, Linear; controlled for baseline levels and performed log transformation of Interferon gamma levels to account for skewed distribution of values; Mean Difference (Final Values) = -16
Statistical Analysis 2: Comparison: Commercially Available Echinacea Product #2 (1 ml/Dose) vs Placebo; Test type: Superiority or Other; p = 0.76, Regression, Linear; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -12

4. Secondary Outcome: Peak Level IL-2
Description: Highest level of IL-2 while taking study medication
Time Frame: 1-10 days after starting study medication
Population: Data analyzed on any participant who IL-2 level was obtained on 1 or more days while on study medication.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Commercially Available Echinacea Product #1 (5 ml/Dose) | Commercially Available Echinacea Product #2 (1 ml/Dose) | Placebo
Number analyzed (Participants) | 22 | 22 | 22
pg/ml | 82 (79) | 148 (321) | 68 (64)
Statistical Analysis 1: Comparison: Commercially Available Echinacea Product #1 (5 ml/Dose) vs Placebo; Test type: Superiority or Other; p = 0.98, Regression, Linear; controlled for baseline levels; Mean Difference (Final Values) = -0.5
Statistical Analysis 2: Comparison: Commercially Available Echinacea Product #2 (1 ml/Dose) vs Placebo; Test type: Superiority or Other; p = 0.34, Regression, Linear; controlled for baseline levels; Mean Difference (Final Values) = 39

5. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Adverse events such as nausea or rash in participants receiving an Echinacea formulation or placebo will be compared
Time Frame: 1- 30 days after starting study medication
Population: Participants who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Commercially Available Echinacea Product #1 (5 ml/Dose) | Commercially Available Echinacea Product #2 (1 ml/Dose) | Placebo
Number analyzed (Participants) | 22 | 22 | 22
participants | 14 | 18 | 16

ADVERSE EVENTS:
Time Frame: day 1 (first dose of study medication) through day 30
Description: Patients specifically inquired about adverse events on day 2, 3, 7, 10, 17 and 30 using 76-item questionnaire.
Arm/Group | Commercially Available Echinacea Product #1 (5 ml/Dose) | Commercially Available Echinacea Product #2 (1 ml/Dose) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 14/22 | 18/22 | 16/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Commercially Available Echinacea Product #1 (5 ml/Dose) (N=22) | Commercially Available Echinacea Product #2 (1 ml/Dose) (N=22) | Placebo (N=22)
Abdominal pain/cramps (Gastrointestinal disorders) | 4 | 3 | 1
Appetite: decreased (Gastrointestinal disorders) | 3 | 1 | 3
Appetite: increased (Gastrointestinal disorders) | 4 | 0 | 1
constipation (Gastrointestinal disorders) | 3 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 3 | 1
Gas/indigestion (Gastrointestinal disorders) | 6 | 3 | 2
Nausea (Gastrointestinal disorders) | 4 | 2 | 2
Thirst: increased (Metabolism and nutrition disorders) | 4 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Headache (Nervous system disorders) | 4 | 5 | 6
Anxiety (Psychiatric disorders) | 3 | 1 | 2
Depression (Psychiatric disorders) | 1 | 1 | 2
Drowsiness/sedation (General disorders) | 3 | 3 | 1
Sleep: excessive (General disorders) | 1 | 3 | 2
Sleep: insomnia, restless (General disorders) | 3 | 4 | 3
Weakness/fatigue (General disorders) | 5 | 4 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 8
Rash/hives (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 4

LIMITATIONS AND CAVEATS:
Levels of TNF alpha, IL-6, IL-2 and Interferon gamma varied widely limiting chance of detecting differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No